CLINICAL TRIAL: NCT04413305
Title: WGS-guided Tracking and Infection Control Measures of Carbapenem-resistant Klebsiella Pneumoniae
Brief Title: WGS-guided Tracking and Infection Control Measures of CRKP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Huashan Hospital (Other)
Collaborators: Sumitomo Pharmaceuticals (Suzhou) Co. Ltd (Unknown)
Responsible Party: Principal Investigator, Wen-hong Zhang, Professor, Huashan Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: KY2019-429KP
Record Dates: First submitted 2020-05-28; First posted 2020-06-02 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: Klebsiella Pneumoniae Infection

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WGS-based screen and control group (Experimental): For intervention group, we screen admitted patients for carbapenem-resistant Klebsiella pneumoniae and carry out 'Bundle' infection and control measures. When outbreak or tranmission of CRKP was observed, we take whole-genome sequencing to track origin and transmission route to decease CRKP rate.
  Interventions: Other: screen of CRKP and infection control measure
- Non-intervention (No Intervention): Non-intervention

INTERVENTIONS:
Other: screen of CRKP and infection control measure — For intervention group, we screen admitted patients for carbapenem-resistant Klebsiella pneumoniae and carry out 'Bundle' infection and control measures. When outbreak or tranmission of CRKP was observed, we take whole-genome sequencing to track origin and transmission route to decease CRKP rate.
  Arms: WGS-based screen and control group

SUMMARY:
The objective of this study is to investigate the effect of the infection control measures based on the active screening of carbapenem-resistant Klebsiella pneumoniae and whole-genome based tracking and surveillance though the hospital.

ELIGIBILITY:
Inclusion Criteria:

1. The patient was admitted to the ICU of neurosurgery in the west hospital of huashan hospital affiliated to fudan university from September 2019 to September 2021, or transferred from the ICU of another hospital
2. The patient is more than 18 years old and less than 80 years old, regardless of gender.
3. Informed consent of the patient;

Exclusion Criteria:

1. Patients participating in other clinical trials at the same time
2. Pregnant

4. People who will affect the outcome of the study: whose specimens could not be received or not enough for testing

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2020-05-28 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Evaluate the influence of WGS-based screen and control measures on the CRKP occurrence rate | 2 years

SECONDARY OUTCOMES:
Analysis of transmission pattern and route pre and post WGS-based tracking | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Infectious department of Huashan Hospital, Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No